CLINICAL TRIAL: NCT01256346
Title: A Comparison of Electrocardiography Versus Pulse Oximetry for Determination of Initial Heart Rate in Preterm Newborns: A Pilot Study.
Brief Title: Electrocardiography Versus Pulse Oximetry for Newborn Heart Rate Determination
Status: Withdrawn | Type: Observational
Why Stopped: Study completed by another institution prior to enrollment of first subject.
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Douglas Dannaway, MD, Assistant Professor of Pediatrics, University of Oklahoma
Other Study IDs: OUHSC IRB 15458
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Prematurity
Keywords: Premature; baby; heart rate; resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Babies: Preterm newborn infants thought to be 24-32 weeks gestational age.
  Interventions: Device: Apparatuses

INTERVENTIONS:
Device: Apparatuses — Each baby will have both pulse oximetry leads (Massimo Radical 7) and electrocardiography leads (3M™ Red Dot™ Neonatal Limb Band Monitoring Electrodes, Pre-wired) applied. The time required for each modality to register a heart rate will be compared.

SUMMARY:
The goal of this study is to compare the time required for accurate heart rate measurement of the preterm newborn when using pulse oximetry versus electrocardiography leads.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 24-32 weeks

Exclusion Criteria:

* Babies with open abdominal defects

Max Age: 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thirty babies believed to be of 24-32 weeks gestational age who are to be born at the University of Oklahoma Health Sciences Center.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time until accurate heart rate. | To be determined
  The elapsed time (in seconds) between application of the specific measuring apparatus (pulse oximeter probe or electrocardiograph leads) and measurement of heart rate.

SECONDARY OUTCOMES:
Intermeasurement accuracy | To be determined
  Assessment of the level of accuracy between the two times to be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dannaway, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Result] Kamlin CO, Dawson JA, O'Donnell CP, Morley CJ, Donath SM, Sekhon J, Davis PG. Accuracy of pulse oximetry measurement of heart rate of newborn infants in the delivery room. J Pediatr. 2008 Jun;152(6):756-60. doi: 10.1016/j.jpeds.2008.01.002. Epub 2008 Mar 6. PMID 18492509
- [Result] Kamlin CO, O'Donnell CP, Everest NJ, Davis PG, Morley CJ. Accuracy of clinical assessment of infant heart rate in the delivery room. Resuscitation. 2006 Dec;71(3):319-21. doi: 10.1016/j.resuscitation.2006.04.015. Epub 2006 Sep 20. PMID 16989935
- [Result] O'Donnell CP, Kamlin CO, Davis PG, Morley CJ. Feasibility of and delay in obtaining pulse oximetry during neonatal resuscitation. J Pediatr. 2005 Nov;147(5):698-9. doi: 10.1016/j.jpeds.2005.07.025. PMID 16291367
- [Result] Owen CJ, Wyllie JP. Determination of heart rate in the baby at birth. Resuscitation. 2004 Feb;60(2):213-7. doi: 10.1016/j.resuscitation.2003.10.002. PMID 15036740
- [Result] Petrozzino JJ, Heldt GP, Rich WD, Finer NN. Use of ECG for initial newborn heart rate assessment: a pilot/feasibility study. J Investig Med. 2008;56(1):263-7.
- [Result] Vento M, Aguar M, Leone TA, Finer NN, Gimeno A, Rich W, Saenz P, Escrig R, Brugada M. Using intensive care technology in the delivery room: a new concept for the resuscitation of extremely preterm neonates. Pediatrics. 2008 Nov;122(5):1113-6. doi: 10.1542/peds.2008-1422. No abstract available. PMID 18977992